CLINICAL TRIAL: NCT02522338
Title: Measurement of Glomerular Filtration Rate (GFR) in HIV Patients: Single-center Study Comparing the Accuracy of Estimators of GFR Versus Iohexol Plasma Clearance
Acronym: HIVOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1008078; 2010-022272-31 (EudraCT Number)
Record Dates: First submitted 2015-08-04; First posted 2015-08-13 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: HIV
MeSH Terms: interventions — Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- iohexol plasma clearance (Other): patients had received iohexol for measuring GFR
  Interventions: Drug: iohexol

INTERVENTIONS:
Drug: iohexol — 10 ml de l'iohexol (300 mgI/ml)

SUMMARY:
Cystatin C, a protease inhibitor produced by most nucleated cells, is freely filtered by the kidneys, and its plasma assay reflects the GFR.

Compare, in HIV patients, the predictive performance of 11 formula to estimate GFR based on assay plasma cystatin C with that of the MDRD formulas.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with HIV, and included in the cohort NADIS

Exclusion Criteria:

* Patient with a known allergy
* Patients treated with metformin
* Patients with severe hepatic impairment defined as a TP spontaneously below 50%
* Patients with a history of dysthyroidism
* Patient with active neoplasia other than skin cancer
* Degradation recent (not older than 3 months) in renal function defined as the deterioration of GFR over 25%.
* Estimated GFR less than 15 mL/min/1, 73m2
* Pregnant or lactating
* Subjects under the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Patient with a predictive performance range -30% to +30% | day 0
  for each estimator :predictive performance calculated by [(DFG estimé* - DFG mesuré par iohexol**)/DFG mesuré par iohexol]X100

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric LUCHT, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France